CLINICAL TRIAL: NCT05374395
Title: Enhancing Substance Use Treatment Services to Decrease Dropout and Improve Outpatient Treatment Utilization in Emerging Adults
Acronym: P2P
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Oregon Social Learning Center (Other); University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Kristyn Zajac, Associate Professor, UConn Health
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-097-2
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Substance Use Disorders
Keywords: peer recovery supports; emerging adults; recovery support services
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomized design will include five blocks of two clinics randomized to the timing of the Peer recovery support-delivered Dropout Prevention enhancement, with each clinic having two phases: a longitudinal Usual Services (US) Phase and a longitudinal Usual Services + Peer recovery support-delivered Dropout Prevention (PDP) enhancement Phase. All clusters will have a baseline phase and will be randomized to the timing of the PDP phase. Once randomized to begin, all clusters will have a 24-month US+PDP Phase.
Who Masked: Outcomes Assessor
Masking Description: Primary outcomes will come from the clinics' chart data. Individuals pulling data from charts will be blind to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Services (No Intervention): clinics will continue to deliver their normal outpatient services
- Peer Recovery Support - Delivered Dropout Prevention + Usual Services (Experimental): clinics will continue to deliver their normal outpatient services plus the peer recovery support-delivered dropout prevention enhancement
  Interventions: Behavioral: Peer Recovery Support-Delivered Dropout Prevention enhancement

INTERVENTIONS:
Behavioral: Peer Recovery Support-Delivered Dropout Prevention enhancement — Peer recovery supports will meet with emerging adults for four weekly sessions plus monthly check-ins during the next two months. Peer recovery supports will engage the emerging adults in motivational and skills-based strategies aimed at increasing adherence to services and attendance to treatment sessions.
  Arms: Peer Recovery Support - Delivered Dropout Prevention + Usual Services

SUMMARY:
Emerging adults (ages 18-25) are at higher risk for substance use disorders, including opiate addiction, than any other age group but are also more likely to drop out early from substance use treatment services. This project will evaluate an enhancement to usual services, delivered by peer recovery supports, specifically aimed at improving treatment adherence and reducing dropout in this age group. The study will also answer key questions about risk factors for dropout among emerging adults and the financial sustainability of enhancing services to reduce dropout.

DETAILED DESCRIPTION:
Emerging adults (EAs; ages 18-25) have higher rates of substance use disorders than any other age group and have been hit particularly hard by the opioid crisis. EAs also demonstrate poor adherence to healthcare regimens associated with substance use services, with higher dropout rates and lower service utilization than any other age group. This poor adherence leads to devastating outcomes, including continued substance use, incarceration, and overdose. In addition, high dropout rates contribute to skyrocketing costs to treatment systems as a result of more acute service needs, expensive service utilization, and long waitlists. Cost-effective strategies that are aimed at improving treatment adherence to substance use services and tailored to meet the unique developmental needs of EAs are an imminent need. Further, little is known about risk factors for dropout specific to this age group, hindering effective system responses to this significant problem.

At the same time, substance use service systems are increasingly using peer recovery supports (PRS; i.e., paraprofessionals who have "lived experience" with substance use problems) to bolster treatment outcomes without incurring considerable additional costs. However, services delivered by PRS have not been tailored specifically to reduce EA dropout, and few have been rigorously tested at all. The current study will evaluate an innovative EA-specific dropout prevention enhancement to usual treatment services, delivered by PRS in community-based substance use treatment clinics (Aim 1). The investigators will employ a stepped-wedge cluster randomized design, resulting in each clinic having a longitudinal usual services phase and a longitudinal dropout prevention phase. The two phases will be compared on rates of EA dropout and service utilization using objective data from clinical charts.

ELIGIBILITY:
Inclusion Criteria:

* 18-25
* initiating outpatient treatment for a substance use problem

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients who dropout from substance use services | 90 days from initiation of treatment
  Data will come from de-identified clinical charts. Dropout will be defined in two ways: 1) patient did not complete the total number of sessions prescribed in the treatment plan and 2) patient was in treatment for less than 90 days.
Number of missed sessions and no show sessions | 90 days from initiation of treatment
  Data will come from de-identified clinical charts. Number of missed sessions or no shows will be evaluated based on the number of scheduled sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Kristyn Zajac, PhD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States